CLINICAL TRIAL: NCT00005052
Title: Adjuvant Ganglioside GM2-KLH/QS-21 Vaccination: Post-Operative Adjuvant Ganglioside GM2-KLH/QS-21 (BMS-248479) Vaccination Treatment After Resection of Primary Cutaneous Melanoma Thicker Than 1.5mm (AJCC/UICC Stage II, T3-T4N0M0), a 2-Arm Multicenter Randomized Phase III Trial vs. Observation
Brief Title: Vaccine Therapy in Treating Patients With Primary Stage II Melanoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067645; EORTC-18961; BMS-CA152-003
Record Dates: First submitted 2000-04-06; First posted 2003-01-27 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2006-01

CONDITIONS: Melanoma (Skin)
Keywords: stage II melanoma
MeSH Terms: conditions — Melanoma | interventions — saponin QA-21V1; Chemotherapy, Adjuvant

INTERVENTIONS:
Biological: GM2-KLH vaccine
Biological: QS21
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. It is not yet known whether vaccine therapy is more effective than observation alone for melanoma.

PURPOSE: This randomized phase III trial is studying vaccine therapy to see how well it works compared to observation alone in treating patients with primary stage II melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effect of immunization with GM2-KLH and QS21 to observation on the disease-free survival of patients with primary cutaneous stage II melanoma after adequate surgery.
* Determine overall survival and toxicity in the two treatment arms.

OUTLINE: This is a randomized, open-label, parallel, multicenter study. Patients are stratified according to participating center, tumor thickness (greater than 1.5 to 3.0 mm vs greater than 3.0 to 4.0 mm vs greater than 4.0 mm), gender, ulceration (yes vs no), and presence of additional staging procedures of regional lymph nodes (yes vs no). Patients are randomized to one of two arms.

* Arm I: Patients are vaccinated with GM2-KLH and QS21 subcutaneously on day 1 of weeks 1-4, 12, 24, 36, 48, 60, 72, 84, 96, 120, and 144 for a total of 14 vaccinations.
* Arm II: Patients undergo observation. Patients are followed every 6 months for 7 years.

PROJECTED ACCRUAL: A total of 1300 patients (650 per arm) will be accrued for this study within 36 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary stage II melanoma greater than 1.5 mm without evidence of lymph node metastases

  * T3 or T4, N0, M0
  * Must originate in the skin
* Wide excision with a minimum of 1-2 cm margin surrounding primary lesion or biopsy scar

  * No more than 56 days since definitive surgical treatment (wide excision)
  * No more than 12 weeks since primary surgery
* No clinical, radiological, or pathological evidence of incompletely resected disease, lymph node metastases, in-transit metastasis, or any distant metastatic disease

PATIENT CHARACTERISTICS:

Age:

* 18 to 80

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.8 g/dL

Hepatic:

* SGOT/SGPT no greater than 2 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2 times ULN
* LDH no greater than 2 times ULN
* Bilirubin no greater than 2 times ULN
* Hepatitis B and C negative

Renal:

* Creatinine normal

Other:

* Not pregnant or nursing
* Negative pregnancy test
* No prior or other concurrent cancer except carcinoma in situ of the cervix or basal or squamous cell skin cancer
* No autoimmune disorders
* No conditions requiring systemic treatment with immunosuppressive drugs including treatment with systemic corticosteroids
* No history of CNS demyelinating or inflammatory disease
* No hereditary or acquired peripheral neuropathy
* No other significant medical or surgical condition or psychiatric disorders requiring medication that would preclude study
* No history of severe allergic reaction to shellfish
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy
* No other concurrent biologic therapy

Chemotherapy:

* No prior systemic chemotherapy
* No concurrent cytotoxic chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy except replacement therapy
* No concurrent corticosteroids
* No concurrent chronic systemic steroids

Radiotherapy:

* No prior adjuvant radiotherapy
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics

Other:

* No prior preoperative infusion or perfusion therapy
* No concurrent immunosuppressive medications
* No other concurrent anticancer therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-12

PRIMARY OUTCOMES:
Disease-free survival

SECONDARY OUTCOMES:
Duration of survival
Toxicity as assessed by CTC v2

CONTACTS AND LOCATIONS:
Overall Officials: Alexander M. M. Eggermont, MD, PhD — Daniel Den Hoed Cancer Center at Erasmus Medical Center
Locations (80):
- Royal Perth Hospital, Perth, Western Australia, Australia
- Belgium (6):
  - Hopital Universitaire Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Hopital de Jolimont, Haine-Saint-Paul
  - U.Z. Gasthuisberg, Leuven
- Denmark (4):
  - Aarhus University Hospital - Aarhus Sygehus - Norrebrogade, Aarhus
  - Rigshospitalet - Copenhagen University Hospital, Copenhagen
  - Herlev Hospital - University Hospital of Copenhagen, Copenhagen
  - Odense University Hospital, Odense
- North-Estonian Regional Hospital Surgical Oncology Centre, Tallinn, Estonia
- Tampere University Hospital, Tampere, Finland
- France (14):
  - CHR de Besancon - Hopital Saint-Jacques, Besançon
  - CHU Ambroise Pare, Boulogne-Billancourt
  - CHU de Caen, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier Regional et Universitaire de Lille, Lille
  - Hopital St. Eloi, Montpellier
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Hopital L'Archet - 2, Nice
  - Hopital Bichat - Claude Bernard, Paris
  - Hopital Saint-Louis, Paris
  - Centre Eugene Marquis, Rennes
  - Centre Hospitalier Regional Metz Thionville, Thionville
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Haematologisch-Onkologische Praxis Altona, Hamburg
  - Universitaets-Hautklinik Wuerzburg, Würzburg
- Israel (2):
  - Rambam Medical Center, Haifa
  - Wolfson Medical Center, Holon
- Italy (10):
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - Ospendale S.M. Annunziata-A.S.DI Florence, Florence
  - Istituto Nazionale per la Ricerca sul Cancro, Genoa (Genova)
  - European Institute of Oncology, Milan
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Milano (Milan)
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Naples
  - Azienda Ospedaliera di Padova, Padua
  - Ospedale S. Camillo-Forlanini, Rome
  - Istituto Regina Elena, Rome
  - Universita Degli Studi di Turin, Torino
- Netherlands (3):
  - Leiden University Medical Center, Leiden
  - Nijmegen Cancer Center at Radboud University Medical Center, Nijmegen
  - Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam
- Norwegian Radium Hospital, Oslo, Norway
- Poland (2):
  - Great Poland Cancer Center, Poznan
  - Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw
- Portugal (2):
  - Instituto Portugues de Oncologia Centro do Porto, S. A., Porto
  - Hospital Distrital De Santarem, Santarém
- Russian Academy of Medical Sciences Cancer Research Center, Moscow, Russia
- Institute of Oncology and Radiology of Serbia, Belgrade, Serbia
- Spain (2):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- United Kingdom (26):
  - Royal Sussex County Hospital, Brighton, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Broomfield Hospital, Chelmsford, Essex, England
  - Cheltenham General Hospital, Cheltenham, England
  - Walsgrave Hospital, Coventry, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Saint Bartholomew's Hospital, London, England
  - Royal Free and University College Medical School, London, England
  - St. George's Hospital, London, England
  - Royal Marsden NHS Foundation Trust - London, London, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - James Cook University Hospital, Middlesbrough, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Poole Hospital NHS Trust, Poole Dorset, England
  - Salisbury District Hospital, Salisbury, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Southend NHS Trust Hospital, Westcliff-on-Sea, England
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Western General Hospital, Edinburgh, Scotland
  - Velindre Cancer Center at Velinde Hospital, Cardiff, Wales
  - Selly Oak Hospital at University Hospital NHS Trust, Birmingham

REFERENCES:
- [Result] Eggermont AM, Suciu S, Ruka W, et al.: EORTC 18961: Post-operative adjuvant ganglioside GM2-KLH21 vaccination treatment vs observation in stage II (T3-T4N0M0) melanoma: 2nd interim analysis led to an early disclosure of the results. [Abstract] J Clin Oncol 26 (Suppl 15): A-9004, 2008.
- [Derived] Patel PM, Suciu S, Mortier L, Kruit WH, Robert C, Schadendorf D, Trefzer U, Punt CJ, Dummer R, Davidson N, Becker J, Conry R, Thompson JA, Hwu WJ, Engelen K, Agarwala SS, Keilholz U, Eggermont AM, Spatz A; EORTC Melanoma Group. Extended schedule, escalated dose temozolomide versus dacarbazine in stage IV melanoma: final results of a randomised phase III study (EORTC 18032). Eur J Cancer. 2011 Jul;47(10):1476-83. doi: 10.1016/j.ejca.2011.04.030. Epub 2011 May 18. PMID 21600759